CLINICAL TRIAL: NCT05007522
Title: Ketotifen and Indomethacin Combination Treatment Clinical Trial for COVID-19 A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Proof-of-Concept Clinical Trial to Evaluate the Efficacy of Ketotifen and Indomethacin for Mild and Moderate COVID-19 in Adults
Brief Title: Ketotifen and Indomethacin Combination Treatment Clinical Trial for COVID-19
Acronym: KICC COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sen-Jam Pharmaceutical (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00108924
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Ketotifen; Indomethacin; ketotifen fumarate ophthalmic solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be provided identical appearing pills
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Drug (Experimental): Ketotifen 2 mg administered in tablet form twice a day (every 12 hr). Indomethacin sustained-release (SR) 75 mg, twice a day (every 12 hr). Patients will be administered 28 doses in total of ketotifen/indomethacin combination.
  Interventions: Drug: Ketotifen/Indomethacin
- Placebo (Placebo Comparator): Placebo pills matching in appearance to study drug twice a day for 28 doses total.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketotifen/Indomethacin — 2 mg tablet, 75 mg SR tablet
  Other Names: Zaditor; Indocin SR; Tivorbex
  Arms: Study Drug
Drug: Placebo — Matching placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of ketotifen and indomethacin taken together to improve symptoms related with COVID-19. Ketotifen and indomethacin are medications approved by the Food and Drug Administration (FDA) to treat diseases other than COVID-19. Their use in this study is investigational, meaning they have not been approved by the FDA to treat COVID-19.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), which is a recently emerged coronavirus that has resulted in an ongoing global pandemic. Fever and cough are most commonly experienced at disease presentation and complications involving the vascular system also occur as potential manifestations of severe disease. In human autopsy studies, infiltration of mononuclear cells in the lung tissue concurrent with edema and hemorrhage are frequently noted5. Other than lung epithelial cells, infection is also observed in endothelial cells, possibly augmenting endothelial activation and vascular permeability6. It is believed that lung pathology during COVID-19 is immune-mediated and compounded by the infiltration of monocytes, neutrophils and subsets of T cells7. Interestingly, perturbations in the numbers of granulocytes in the blood, such as neutrophils and eosinophils have also been shown to be associated with severe disease1, 8, 9.

Mast cells (MCs) are long-lived granulated immune cells that are present in both connective and mucosal tissues10. Our data in animal models support that MCs are strongly activated during infection by SARS-CoV-2 virus. Animal studies suggested that drugs in the class of MC "stabilizers" can effectively limit vascular leakage in mouse models of viral infection, such as caused by dengue virus (DENV).

Ketotifen is an oral drug currently used to prevent asthma. It is used to treat irritation and reduce vascular leakage, such as in the eye. It is a MC stabilizing agent that prevents degranulation of MCs, as well as the production of additional mediators that are not contained within MC granules, including leukotrienes and platelet activating factor 32. Indomethacin is an inhibitor of cyclooxygenase (COX) 1 and 2 receptors and, therefore, its primary mechanism of action is through inhibition of prostaglandin synthesis. It is used to treat inflammatory disorders and pain including rheumatoid arthritis, tendinitis, gout, and nephrogenic diabetes insipidus due to its antipyretic and analgesic properties.

This is a randomized, double blind, placebo-controlled, clinical study of ketotifen and indomethacin in adults 18 to 75 years of age, who meet at least two symptoms indicating COVID-19 infection, and who test positive for COVID-19 infection by a PCR based assay or rapid detection assay. Patients meeting all inclusion and exclusion criteria will be enrolled. Eligible patients who present at or are referred to trial sites will undergo screening. Trained research staff will obtain informed consent from participants. Patients meeting all inclusion and exclusion criteria and who agree to participate will be enrolled for the duration of the study.The study will be conducted as an outpatient study. One hundred and fifty (150) patients will be randomized 2:1 to ketotifen/indomethacin or placebo.

The primary objectives is as follows:

To evaluate the safety ketotifen and indomethacin, in combination, in COVID-19 patients.

Hypothesis: This drug combination will be safe in COVID-19 patients, with no increase in adverse events, and no increased severity of COVID-19 disease. (clinical endpoint)

To investigate the effectiveness of ketotifen and indomethacin for improving clinical measures of respiratory function and/or resolution of COVID-19 symptoms.

Hypothesis: Combination treatment of COVID-19 patients with ketotifen and indomethacin will improve patient measures of shortness of breath and/or promote the resolution of COVID-19 respiratory symptoms, shortening the duration of those symptoms. (clinical endpoint)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-75 years
2. Has SARS-CoV-2-positive antigen or molecular diagnostic test (validated SARS-CoV-2 antigen, RT-PCR, or other molecular diagnostic assay from a sample collected no more than 7 days prior to enrollment.
3. At least two signs or symptoms of disease consistent with acute COVID-19 infection. One of these two symptoms must include cough OR shortness of breath with onset within 7 days prior to randomization. Other symptoms that qualify include:

   1. Fever
   2. nausea
   3. vomiting
   4. diarrhea
   5. muscle aches
   6. fatigue
   7. headache
   8. loss of smell or taste
   9. others that are consistent with acute COVID-19 infection in the opinion of the Investigator.
4. Able and willing to give written or oral informed consent
5. Willing to be an outpatient from Study Day 1 to 14, to provide blood during patient visits on Study Days 1, 3, 5, and 10, return on Study Days 1, 3, 5, 7, 10, 14, and 21 for assessment.
6. Willing to keep a diary of pain medication usage, side effects, and COVID-19 associated symptoms and answer a follow-up questionnaire on Study Day 84.

Exclusion Criteria:

1. Clinical signs and symptoms for severe COVID-19, such as:

   1. Need for hospitalization at the time of screening
   2. Need for supplemental O2 at the time of screening
2. A person with any of the following laboratory values:

   1. AST or ALT >/= 1000 U/L
   2. Known serum creatinine > 1.6 mg/dL
3. Prior use of any of the following treatments: COVID-19 convalescent plasma, monoclonal antibodies against SARS-CoV-2, IVIG (for COVID-19), or COVID-19 treatments (authorized, approved, or investigational)
4. Current usage (within the last 7 days prior to randomization) of any of the following drugs:

   1. anticoagulant drugs including, but not limited to, aspirin, warfarin, or clopidogrel.
   2. systemic corticosteroids or non-steroidal anti-inflammatory medications for any indication
   3. drugs that are known to block the functions of ketotifen, such as propranolol.
   4. oral anti-diabetic agents
   5. diflunisal or other drugs (or drugs at certain doses) that are contraindicated for concurrent use with Indomethacin
5. Prior vaccination of at least one dose of vaccine for SARS-CoV-2
6. Has participated, is participating, or plans to participate in a clinical research study evaluating any authorized, approved, or investigational drug SARS-CoV-2
7. Any other clinically significant acute illness within 7 days prior to first study drug administration that would impact outcome assessment.
8. Patients with a history of any gastrointestinal bleeding requiring medical care.
9. Exposure to any new investigational agent within 30 days prior to the study drug administration.
10. Clinically significant abnormal physical examination unrelated to COVID-19 infection that would impact outcome assessment.
11. Females who are pregnant or breast feeding.
12. Current significant medical condition or illness including cardiac arrhythmias, cardiomyopathy or other cardiac disease, advanced renal disease, immunocompromised state including known HIV infection, or any other illness that the Investigator considers should exclude the patient, especially those that require continuation of other medications likely to have an interaction with the study drug. Patients with a history of allergy will not be excluded unless the allergy may be directed to the Study Drug, other NSAIDs, or other tablet ingredient.
13. Any condition that would render the informed consent invalid, or limit the ability of the patient to comply with the study requirements.
14. Inability to comply with completing the outcome assessment measure(s).
15. Any condition that, in the opinion of the investigator, would complicate or compromise the study or well-being of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
UCSD Shortness of Breath Questionnaire | Study Day 14
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.

SECONDARY OUTCOMES:
Development of severe disease | 28 days
  Severe disease defined as hypoxia to room air pulse oximetry below 93%
Development of severe disease | 84 days
  Severe disease defined as hypoxia to room air pulse oximetry below 93%
Development of severe disease | 14 days
  Severe disease defined as hypoxia to room air pulse oximetry below 93%
Proportion and number of medically attended visits related to COVID-19 | 28 days
  Need for emergency department visit or hospitalization for symptoms of COVID-19
Proportion and number of medically attended visits related to COVID-19 | 84 days
  Need for emergency department visit or hospitalization for symptoms of COVID-19
Need for hospitalization | 28 days
  inpatient hospitalization
Need for hospitalization | 84 days
  inpatient hospitalization
Intensive care unit admission | 28 days
  Intensive care unit admission
Intensive care unit admission | 84 days
  Intensive care unit admission
Supplemental oxygen | 28 days
  Clinical care provider prescribing supplemental oxygen
Supplemental oxygen | 84 days
  Clinical care provider prescribing supplemental oxygen
Need for mechanical ventilation | 28 days
  Clinical care provider prescribing mechanical ventilation
Need for mechanical ventilation | 84 days
  Clinical care provider prescribing mechanical ventilation
severe functional disability (WHO ordinal scale) | 28 days
  WHO Ordinal Scale
severe functional disability (WHO ordinal scale) | 84 days
  WHO Ordinal Scale
UCSD Shortness of Breath Questionnaire | Day 84
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 2
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 3
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 4
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 5
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 6
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 7
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 8
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 9
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 10
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 11
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 12
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
UCSD Shortness of Breath Questionnaire | Day 13
  24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living.
Serum chymase concentration | day 10
  Serum chymase concentration
Serum chymase concentration | day 5
  Serum chymase concentration
Serum chymase concentration | day 3
  Serum chymase concentration
coagulation | day 3
  Hematocrit, platelets, PT/PTT
coagulation | day 5
  Hematocrit, platelets, PT/PTT
coagulation | day 10
  Hematocrit, platelets, PT/PTT
Patient Global Improvement Score | Day 14
  A questionnaire that results in a numerical value that is the sum of the patients responses to questions on a likert scale
Patient Global Improvement Score | Day 84
  A questionnaire that results in a numerical value that is the sum of the patients responses to questions on a likert scale
Patient Global Improvement Score | Day 28
  A questionnaire that results in a numerical value that is the sum of the patients responses to questions on a likert scale
Incidence of associated symptoms of COVID-19 | Day 14
  Incidence of symptoms associated with allergy, respiratory viral infection, and/or vascular pathology
Incidence of associated symptoms of COVID-19 | Day 28
  Incidence of symptoms associated with allergy, respiratory viral infection, and/or vascular pathology
Incidence of associated symptoms of COVID-19 | Day 84
  Incidence of symptoms associated with allergy, respiratory viral infection, and/or vascular pathology
adverse effect profile | Day 14
  incidence of GI upset, ulcers, and renal function
adverse effect profile | Day 28
  incidence of GI upset, ulcers, and renal function
adverse effect profile | Day 84
  incidence of GI upset, ulcers, and renal function

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Limkakeng, MD, Principal Investigator — Duke University
Locations (2):
- Nepal (2):
  - Dhulikhel Hospital, Kavre, Bagmati
  - Global Clinical Research Pvt. Ltd., Kathmandu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St John AL, Rathore APS. Early Insights into Immune Responses during COVID-19. J Immunol. 2020 Aug 1;205(3):555-564. doi: 10.4049/jimmunol.2000526. Epub 2020 Jun 8. PMID 32513850
- [Background] Abraham SN, St John AL. Mast cell-orchestrated immunity to pathogens. Nat Rev Immunol. 2010 Jun;10(6):440-52. doi: 10.1038/nri2782. PMID 20498670
- [Background] St John AL, Abraham SN. Innate immunity and its regulation by mast cells. J Immunol. 2013 May 1;190(9):4458-63. doi: 10.4049/jimmunol.1203420. PMID 23606723
- [Background] Rathore AP, St John AL. Protective and pathogenic roles for mast cells during viral infections. Curr Opin Immunol. 2020 Oct;66:74-81. doi: 10.1016/j.coi.2020.05.003. Epub 2020 Jun 18. PMID 32563779
- [Background] Kiani P, Scholey A, Dahl TA, McMann L, Iversen JM, Verster JC. In Vitro Assessment of the Antiviral Activity of Ketotifen, Indomethacin and Naproxen, Alone and in Combination, against SARS-CoV-2. Viruses. 2021 Mar 26;13(4):558. doi: 10.3390/v13040558. PMID 33810356